CLINICAL TRIAL: NCT07071467
Title: Innovative Clean-Seal Technique Incorporating Sodium Hypochlorite and Hyaluronic Acid as an Adjunct to Non-Invasive Therapy for Stage III Periodontitis Management
Brief Title: Testing Sodium Hypochlorite and Hyaluronic Acid as an Adjunct to Non-Invasive Therapy for Stage III Periodontitis Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karim Ismail (Other)
Responsible Party: Sponsor-Investigator, Karim Ismail, MSc. candidate in the diagnosis, oral medicine & periodontology department, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 9208891
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Periodontitis (Stage 3); Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing; Sodium Hypochlorite; Hyaluronic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scaling and root planing with sodium hypochlorite and hyaluronic acid (Experimental)
  Interventions: Other: Scaling and root planing with sodium hypochlorite and hyaluronic acid
- Scaling and root planing (Active Comparator)
  Interventions: Procedure: Scaling and root planing

INTERVENTIONS:
Other: Scaling and root planing with sodium hypochlorite and hyaluronic acid — Sodium hypochlorite gel was applied first for 30 seconds, then followed by subgingival instrumentation of the site. Then, 1.8% hyaluronic acid (1.6% cross-linked, 0.2% natural hyaluronic acid ) was applied subgingivally into the periodontal pocket to seal the site.
  Arms: Scaling and root planing with sodium hypochlorite and hyaluronic acid
Procedure: Scaling and root planing — Pockets were treated with sub-gingival scalling and root planning alone.
  Arms: Scaling and root planing

SUMMARY:
The study was designed to evaluate the concept of the clean & seal, using sodium hypochlorite gel and hyaluronic acid as adjunctive to non-surgical therapy for management of Stage III Periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes diagnosed with periodontitis Stage III.
* CAL ≥ 5mm or bone loss affecting middle third of the root in more than two adjacent teeth.
* PPD ≥ 6mm in more than two adjacent teeth.
* Periodontal tooth loss ≤ 4 teeth.
* Systemically healthy patients.

Exclusion Criteria:

* Patient with uncontrolled diabetes.
* Pregnant or lactating.
* Tobacco smoker ≥ 10 cigarettes/day.
* Antibiotic treatment within previous 4 weeks.
* Acute periodontal or periapical abscess

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Plaque accumulation | up to 12 weeks
  This was assessed using O'Leary plaque index. The O'Leary Plaque Index records the presence or absence of dental plaque on four surfaces (mesial, distal, buccal, lingual) of each tooth. The score ranges from 0% (no plaque) to 100% (plaque on all surfaces), with lower percentages indicating better oral hygiene.
Gingival condition assessment | up to 12 weeks
  The Gingival Index of Löe and Silness was used to assess the severity of gingival inflammation based on color, consistency, and bleeding on probing across four areas per tooth. Scores range from 0 (normal gingiva) to 3 (severe inflammation with spontaneous bleeding), with higher scores indicating worse gingival health.

SECONDARY OUTCOMES:
Probing depth | up to 12 weeks
  Probing Depth is the measurement of the distance from the gingival margin to the bottom of the periodontal pocket using a periodontal probe. Values typically range from 1-3 mm (healthy) to ≥5 mm (indicative of periodontal disease), with deeper pockets reflecting more severe attachment loss.
Clinical attachment loss | up to 12 weeks
  Clinical Attachment Loss measures the distance from the cementoenamel junction to the base of the periodontal pocket, indicating the extent of periodontal support lost. Values range from 0 mm (no attachment loss) to ≥5 mm or more (severe loss), with higher measurements reflecting greater periodontal destruction.

OTHER OUTCOMES:
Microbiological assessment of P. gingivalis | 6 weeks
  The bacteriological parameter by using Real Time PCR was used to evaluate the Porphyromonas gingivalis load.
  Sub-gingival plaque samples were taken by removing of the supra-gingival plaque with curette and cotton pellets before inserting , sterile endodontic paper points in periodontal pocket and leaving them in situ for 10 seconds. The paper points were immediately transferred to sterile , dry cryovials . Paper points were stored frozen at -80 ºC immediately after sample collection until being processed with PCR.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt